CLINICAL TRIAL: NCT02745691
Title: An International Phase 4 Field Study for Analyzing the Psychometric Properties of the Updated Module on Assessing Quality of Life of Patients With Lung Cancer (EORTC QLQ-LC29)
Brief Title: Psychometric Properties of the EORTC QLQ-LC29
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Michael Koller, Head, Center of Clinical Studies, University Hospital Regensburg
Other Study IDs: LC29_Phase4
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: quality of life; psychometric validation; international field study; patient-reported outcome (PRO)
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative; Chemoradiotherapy; Bevacizumab; Erlotinib Hydrochloride; Gefitinib; Crizotinib; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A. Surgery: A.1 Surgery alone and/or before any adjuvant therapy A.2 Surgery (late effects)
  Interventions: Other: Surgery
- B. Radiochemotherapy: B.1 Chemotherapy alone B.2 Radiotherapy alone B.3 Sequential radiochemotherapy B.4 Concurrent radiochemotherapy
  Interventions: Other: Radiochemotherapy
- C. Targeted therapy: C.1 Targeted therapy alone C.2 Targeted therapy in combination with any other therapy
  Interventions: Other: Targeted therapy
- D. Immunotherapy: Any new immunotherapy for lung cancer
  Interventions: Other: Immunotherapy

INTERVENTIONS:
Other: Surgery — Thoracic surgery for lung cancer
  Groups: A. Surgery
Other: Radiochemotherapy — Either chemotherapy or radiotherapy alone or combination of both (either subsequent or concurrent)
  Groups: B. Radiochemotherapy
Other: Targeted therapy — New targeted therapies for lung cancer
  Other Names: Bevacizumab, Erlotinib, Gefitinib, and Crizotinib
  Groups: C. Targeted therapy
Other: Immunotherapy — New immunotherapies for lung cancer
  Groups: D. Immunotherapy

SUMMARY:
The aim of the Phase 4 study is to test the scale structure, reliability, responsiveness to change and validity of the EORTC QLQ-LC29 in conjunction with the EORTC QLQ-C30 in patients diagnosed with lung cancer. Participants will be enrolled in four groups according to their primary therapy (A. Surgery, B. Radiochemotherapy, C. Targeted therapy, D. Immunotherapy). According to sample size calculations the investigators will include a total of N = 450 patients, but inflating the recruitment goal is permissible.

DETAILED DESCRIPTION:
Background The EORTC QLQ-C30 assesses quality of life of cancer patients and comprises 30 items that are grouped in five functional scales (physical, role, cognitive, emotional and social), one scale to rate global health and quality of life, three multi-item symptom scales (fatigue, nausea and vomiting, pain) and five single symptom items (dyspnoea, insomnia, appetite loss, constipation and diarrhea), one item assessing perceived financial impact of disease and treatment.

The updated lung cancer module, the QLQ-LC29, is a module to be used in conjunction with the QLQ-C30 for the assessment of specific aspects of quality of life in patients with lung cancer. All items are accompanied by the classic EORTC four-point Likert response scale with the labels 1 "not at all", 2 "a little", 3 "quite a bit", and 4 "very much". The time frame is the past week ("Please indicate the extent to which you have experienced these symptoms or problems during the past week").

Eligibility Patients are eligible for this study if they have a histologically confirmed diagnosis of lung cancer, are able to understand the language of the questionnaire, are mentally fit to complete the questionnaire, and have provided written informed consent.

Sampling matrix Participants will be enrolled in four groups according to their primary therapy: A. Surgery, B. Radiochemotherapy, C. Targeted therapy, D. Immunotherapy. Various combinations of therapies are possible, resulting in a total of eight subgroups: A.1 Surgery alone and/or before any adjuvant therapy, A.2 Surgery (late effects), B.1 Chemotherapy alone, B.2 Radiotherapy alone, B.3 Sequential radiochemotherapy, B.4 Concurrent radiochemotherapy, C.1 Targeted therapy alone, C.2 Targeted therapy in combination with any other therapy, D. Immunotherapy.

Procedure Patients are informed about the goal of the study. After granting informed consent, patients fill in the self-administered paper version of the EORTC QLQ-C30 plus the new lung module QLQ-LC29. Their physicians provide the clinical documentation. A subsample of the patients will fill in the questionnaires at a second time point two to four weeks later.

Sample size According to sample size calculations we will include a total of N = 450 patients, but inflating the recruitment goal is permissible.

Statistical analyses Scale structure will be analysed by confirmatory factor analyses, and backed by classical test theory (convergent/discriminant validity). Reliability will be calculated by means of Cronbach's alpha (internal consistency) and intra-class coefficient (ICC, test-retest reliability). Sensitivity of the module will be assessed by means of known group differences (Karnofsky Performance Status). Responsiveness to change over time will take into account differences between the second and first assessment.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of lung cancer
* no previous primary or recurrent tumour
* ability to understand the language of the questionnaire
* mental fitness to complete a questionnaire
* 18 years of age or above
* written informed consent.-

Exclusion Criteria:

* no histologically confirmed diagnosis of lung cancer-
* previous primary or recurrent tumour
* not mentally fit to complete a questionnaire
* not able to understand the language of the questionnaire
* younger than 18
* refusal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed diagnosis of lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
QLQ-LC29 | In the course of therapy or up to three months after having completed therapy
  Self-reported symptoms related to lung cancer. Each item is rated on a response scale 1 = not at all to 4 = very much and refer to the time frame "during the past week"

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koller, PhD, Principal Investigator — University Hospital Regensburg
Locations (1):
- Center for Clinical Studies, University Hospital Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch M, Grafenstein L, Karnosky J, Schulz C, Koller M. Psychosocial Burden and Quality of Life of Lung Cancer Patients: Results of the EORTC QLQ-C30/QLQ-LC29 Questionnaire and Hornheide Screening Instrument. Cancer Manag Res. 2021 Aug 7;13:6191-6197. doi: 10.2147/CMAR.S314310. eCollection 2021. PMID 34393512
- [Derived] Koller M, Shamieh O, Hjermstad MJ, Hornslien K, Young T, Chalk T, Ioannidis G, Harle A, Johnson CD, Tomaszewski KA, Serpentini S, Pinto M, van der Weijst L, Janssens A, Morag O, Chie WC, Arraras JI, Pompili C, Jungraithmayr W, Hechtner M, Katsochi D, Muller K, Grafenstein L, Schulz C, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group; EORTC Lung Cancer Group; European Society of Thoracic Surgeons. Psychometric properties of the updated EORTC module for assessing quality of life in patients with lung cancer (QLQ-LC29): an international, observational field study. Lancet Oncol. 2020 May;21(5):723-732. doi: 10.1016/S1470-2045(20)30093-0. Epub 2020 Mar 23. PMID 32213338